CLINICAL TRIAL: NCT01681277
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Doses of BI 113608 Powder for Oral Solution in Healthy Male Volunteers q.d. or b.i.d. for 14 Days (a Randomised, Double-blind, Placebo-controlled Within Dose Groups Phase I Trial)
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Doses of BI 113608 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1314.2; 2012-002536-82 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2016-11

CONDITIONS: Healthy

ARMS (4):
- BI 113608 high dose bid (Experimental): powder in the bottle for oral solution, oral administration with 240 ml water
  Interventions: Drug: Placebo to BI 113608 PIB bid; Drug: BI 113608 PIB bid
- BI 113608 low dose bid (Experimental): powder in the bottle for oral solution, oral administration with 240 ml water
  Interventions: Drug: Placebo to BI 113608 PIB bid; Drug: BI 113608 PIB bid
- BI 113608 medium dose bid (Experimental): powder in the bottle for oral solution, oral administration with 240 ml water
  Interventions: Drug: BI 113608 PIB bid; Drug: Placebo to BI 113608 PIB bid
- BI 113608 high dose qd (Experimental): powder in the bottle for oral solution, oral administration with 240 ml water
  Interventions: Drug: Placebo to BI 113608 PIB qd; Drug: BI 113608 PIB qd

INTERVENTIONS:
Drug: BI 113608 PIB bid — powder for oral solution
  Arms: BI 113608 medium dose bid
Drug: Placebo to BI 113608 PIB bid — powder for oral solution
  Arms: BI 113608 low dose bid
Drug: Placebo to BI 113608 PIB bid — powder for oral solution
  Arms: BI 113608 medium dose bid
Drug: Placebo to BI 113608 PIB qd — powder for oral solution
  Arms: BI 113608 high dose qd
Drug: Placebo to BI 113608 PIB bid — powder for oral solution
  Arms: BI 113608 high dose bid
Drug: BI 113608 PIB bid — powder for oral solution
  Arms: BI 113608 high dose bid
Drug: BI 113608 PIB bid — powder for oral solution
  Arms: BI 113608 low dose bid
Drug: BI 113608 PIB qd — powder for oral solution
  Arms: BI 113608 high dose qd

SUMMARY:
The objective of the current trial is to evaluate safety, tolerability and pharmacokinetics of multiple rising doses of BI 113608 in healthy male volunteers

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects were orally administered matching placebo to BI 113608 (powder in the bottle for oral solution) with 240 ml water after an overnight fast of at least 10 h. Subjects were treated for 14 days. Each subject received a single morning dose on Day 1 and Day 14 for all dose group, twice daily dose (b.i.d.) on Days 2 to 13 for dose group 1 to 3 and a single morning dose (q.d.) for group 4.
- BI 113608 25 mg Bid (DG1): Dose Group (DG) 1: Subjects were orally administered with daily dose of BI 113608 50 mg (25 mg b.i.d) (powder in the bottle for oral solution) with 240 ml water after an overnight fast of at least 10 h. Subjects were treated for 14 days. Each subject received a single morning dose on Day 1, followed by a 12-days (b.i.d. treatment on Days 2 to 13, and a single morning dose on Day 14.
- BI 113608 50 mg Bid (DG2): DG 2: Subjects were orally administered with daily dose of BI 113608 100 mg (50 mg b.i.d) (powder in the bottle for oral solution) with 240 ml water after an overnight fast of at least 10 h. Subjects were treated for 14 days. Each subject received a single morning dose on Day 1, followed by a 12-days b.i.d. treatment on Days 2 to 13, and a single morning dose on Day 14.
- BI 113608 100 mg Bid (DG3): DG 3: Subjects were orally administered with daily dose of BI 113608 200 mg (100 mg b.i.d) (powder in the bottle for oral solution) with 240 ml water after an overnight fast of at least 10 h. Subjects were treated for 14 days. Each subject received a single morning dose on Day 1, followed by a 12-days b.i.d. treatment on Days 2 to 13, and a single morning dose on Day 14.
- BI 113608 100 mg qd (DG4): DG 4: Subjects were orally administered with daily dose of BI 113608 100 mg (100 mg q.d) (powder in the bottle for oral solution) with 240 ml water after an overnight fast of at least 10 h. Subjects were treated for 14 days. Each subject received a single morning dose on Day 1 to Day 14.
Period: Overall Study
Arm/Group | Placebo | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Started | 12 | 9 | 9 | 9 | 9
Completed | 11 | 9 | 9 | 9 | 9
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This set included all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug. The TS included all 48 treated subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4) | Total
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (7.0) | 40.9 (7.0) | 44.2 (5.7) | 43.8 (4.6) | 40.1 (8.0) | 41.9 (6.5)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 12 | 9 | 9 | 9 | 9 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentage of participants with drug-related adverse events
Time Frame: From administration of study drug until end-of-study, up to 17 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
percentage of participants | 33.3 | 33.3 | 22.2 | 88.9 | 77.8

2. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities for Clinical Laboratory Evaluation, Vital Signs, and ECG Recordings
Description: Number of participants with Clinically relevant abnormalities for clinical laboratory tests (haematology, clinical chemistry and urinalysis), vital signs (blood pressure (BP), pulse rate (PR), respiratory rate (RR), body temperature), and 12- lead electrocardiogram (ECG)
Time Frame: From administration of study drug until end-of-study, up to 17 days
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Placebo | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 12 | 9 | 9 | 9 | 9
participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Cmax,ss
Description: Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss).
Time Frame: 311.917h before dose and 312.25h. 312.5h, 312.75h, 313h, 313.5h, 314h, 314.5h, 315h, 316h, 318h, 320h, 322h, 324h, 328h, 336h after last dose. The time 324h for the b.i.d treatment and 336h for the q.d. treatment.
Population: PK analysis set (PKS): This set included all subjects of the TS who provided at least one observation for at least one secondary PK endpoint without important protocol violations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 9 | 9 | 9 | 9
nmol/L | 119 (58.2) | 261 (40.3) | 648 (27.7) | 549 (41.7)
Statistical Analysis 1: Comparison: BI 113608 25 mg Bid (DG1) vs BI 113608 50 mg Bid (DG2) vs BI 113608 100 mg Bid (DG3) vs BI 113608 100 mg qd (DG4); This was non confirmatory testing (Single dose). Dose proportionality of BI 113608 for Cmax,ss was analysed; Test type: Superiority or Other; Slope = 1.2208, 95% CI 2-sided [0.9354 to 1.5062], Standard Error of Mean 0.1386 — Dose proportionality was explored using the power model (ANCOVA). The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale. Standard Error of the mean is actually the Standard Error of the slope

4. Secondary Outcome: Tmax,ss
Description: Time from last dosing to maximum concentration of the analyte in plasma at steady state (tmax,ss).
Time Frame: as for outcome 3
Population: PKS
Measure: Median (Full Range); unit: h
Arm/Group | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 9 | 9 | 9 | 9
h | 0.500 [0.250 to 0.500] | 0.500 [0.250 to 2.00] | 0.750 [0.500 to 1.00] | 0.750 [0.250 to 4.00]

5. Secondary Outcome: AUCtau,ss
Description: Area under the concentration-time curve of the analyte BI 113608 in plasma at steady state over a uniform dosing interval t (AUCtau,ss).
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 9 | 9 | 9 | 9
nmol*h/L | 491 (48.5) | 1290 (29.0) | 3030 (32.2) | 2290 (20.0)
Statistical Analysis 1: Comparison: BI 113608 25 mg Bid (DG1) vs BI 113608 50 mg Bid (DG2) vs BI 113608 100 mg Bid (DG3) vs BI 113608 100 mg qd (DG4); This was non confirmatory testing (Single dose). Dose proportionality of BI 113608 for AUCt,ss was analysed; Test type: Superiority or Other; Slope = 1.3135, 95% CI 2-sided [1.0652 to 1.5618], Standard Error of Mean 0.1206 — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: t1/2,ss
Description: Terminal half-life of the analyte in plasma at steady state (t1/2,ss).
Time Frame: 311.917h before dose and 312.25h. 312.5h, 312.75h, 313h, 313.5h, 314h, 314.5h, 315h, 316h, 318h, 320h, 322h, 324h, 328h, 336h, 360h, 384h after last dose.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 9 | 9 | 9 | 9
h | 14.0 (15.4) | 12.9 (22.8) | 12.9 (14.7) | 13.1 (15.6)

7. Secondary Outcome: RA,Cmax
Description: Accumulation ratio of the analyte in plasma at steady state after multiple oral administration over a uniform dosing interval t, expressed as ratio of Cmax at steady state and after single dose (RA,Cmax).
Time Frame: -2h,0.25h,0.5h,0.75h,1h,1.5h,2h,2.5h,3h,4h,6h,8h,10h,12h,16h,23.917h and 311.917h before dose and 312.25h. 312.5h, 312.75h, 313h, 313.5h, 314h, 314.5h, 315h, 316h, 318h, 320h, 322h, 324h, 328h, 336h after single and multiple dose.
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Ratio | 1.36 (54.0) | 1.15 (23.6) | 1.09 (34.3) | 0.915 (38.8)

8. Secondary Outcome: RA,AUC
Description: Accumulation ratio of the analyte in plasma at steady state after multiple dose administration over a uniform dosing interval t, expressed as ratio of AUC at steady state and after single dose (RA,AUC).
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Ratio | 1.29 (29.9) | 1.48 (13.0) | 1.37 (14.5) | 1.05 (15.6)

ADVERSE EVENTS:
Time Frame: From administration of study drug until end-of-study, up to 17 days
Arm/Group | Placebo | BI 113608 25 mg Bid (DG1) | BI 113608 50 mg Bid (DG2) | BI 113608 100 mg Bid (DG3) | BI 113608 100 mg qd (DG4)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 5/12 | 4/9 | 2/9 | 8/9 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | BI 113608 25 mg Bid (DG1) (N=9) | BI 113608 50 mg Bid (DG2) (N=9) | BI 113608 100 mg Bid (DG3) (N=9) | BI 113608 100 mg qd (DG4) (N=9)
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 8 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 5 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 0
Feeling of relaxation (General disorders) | 0 | 0 | 0 | 1 | 0
Sensation of pressure (General disorders) | 0 | 0 | 0 | 1 | 0
Spinal pain (General disorders) | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.